CLINICAL TRIAL: NCT06548022
Title: Rare Group Problem Management Plus
Acronym: Group PM+
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: Travere Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Maureen Lyon, Clinical Health Psychologist, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRBear Protocol # 1049
Record Dates: First submitted 2024-07-29; First posted 2024-08-12 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Anxiety; Depressive Symptoms; Post-traumatic Stress Disorder; Problems Psychosocial
Keywords: rare disease; pediatric; family caregiver; psychoeducation; group intervention
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic; Rare Diseases

STUDY DESIGN:
Intervention Model Description: Single group, pre/post-test design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rare Group PM Plus (Experimental): Rare Group PM Plus consists of 5 weekly sessions. Each session lasts 90 minutes.
  Session 1: Managing Stress Session 2: Managing Problems Session 3: Get Going, Keep Doing Session 4: Strengthening Social Support Session 5: Staying Well and Looking Forward
  Interventions: Behavioral: Rare Group Problem Management Plus

INTERVENTIONS:
Behavioral: Rare Group Problem Management Plus — The World Health Organization's Group Problem Management Plus (Group PM+) intervention has been demonstrated to effectively provide psychological help for adults impaired by distress in communities exposed to adversity. Investigators will test an adapted model for use on-line and with family caregivers of children with rare diseases. Managing Stress. Teaching participants a brief stress management strategy will help them better manage problems related to anxiety and stress. Managing Problems. This is a strategy to apply in situations where a participant is experiencing practical problems (e.g. conflict in the family). Get Going, Keep Doing. This strategy targets depression and inactivity. Strengthening Social Support. Individuals with emotional problems can be isolated from supportive people and organizations. Strengthening social support promotes well-being. Staying Well and Looking Forward. This is a review, ends with a closing ceremony.

SUMMARY:
Participants are being asked to be in the study if they are the parent or legal guardian of a child (>1 year or <18 years old) with a rare condition.

The group based psychoeducational intervention is called Rare Group Problem Management Plus.

Rare Group PM Plus may help adults with practical and emotional problems. It is a group program (there will be other men or women with similar problems) It happens once a week for 5 weeks (each session lasts 90 minutes)

Participants will complete assessments before they start Rare Group PM+. Participants will also complete the same assessments within a few weeks of completing Rare Group PM+. Assessments should only take one hour.

Study visits are by Telemedicine. Participants will need a smart phone or tablet. If they do not have a smart phone or tablet, the study team will help with this.

Participants will not receive any materials or money or medication.

DETAILED DESCRIPTION:
Participants are being asked to be in the study because they are the parent or legal guardian of a child (infancy up to 21 years old) with a rare condition.

The group based psychoeducational intervention is called Rare Group Problem Management (PM) Plus intervention.

Rare Group PM Plus may help adults with practical and emotional problems It is a group program (there will be other men or women with similar problems) It happens once a week for 5 weeks (each session lasts 90 minutes)

Investigators will be recruiting for 3 groups of 10 families each, for a total of 30 families who will participate in this study from Children's National Hospital.

There are 7 study visits.

Study Timeline:

Study visit 1: Assessment-Before Group PM+ Study visit 2: Session 1-Managing Stress Study visit 3: Session 2-Managing Problems Study visit 4: Session 3-Get Going, Keep Doing Study visit 5: Session 4-Strengthening Social Support Study Visit 6: Session 5-Staying Well and Looking Forward Study Visit 7: Assessment within 2 weeks after complete Group PM+

Sessions will occur over Zoom Telehealth and facilitated by a licensed clinical psychologist and a genetic counselor trainee.

Investigators will use chi-square tests and Fisher's exact test to measure changes from baseline to 2 weeks post-intervention. Investigators will also collect qualitative data on what participants liked about the intervention, what they did not like, and what they think will improve the intervention.

ELIGIBILITY:
Inclusion Criteria:

* • Family caregiver aged 18 years or older of a child with a rare disease from infancy to age 21 years.

  * Understands and speaks English or Spanish. Reading or health literacy is not required.
  * Signed consent.
  * Signed waiver of assent for child.

Exclusion Criteria:

* Family caregiver is under the age of 18 years.
* Child with the rare disease is over the age of 21 years.
* Family caregiver is actively suicidal, homicidal, or psychotic.
* Family caregiver is impaired (cognitively or by drugs or alcohol).
* Family caregiver has a low level of distress.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability | 2 weeks post-intervention (Session 5)
  As measured by retention at 2 weeks post-intervention assessment

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Lyon, PhD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available to other researchers for this development and adaptation study.

REFERENCES:
- [Background] Bogart KR, Irvin VL. Health-related quality of life among adults with diverse rare disorders. Orphanet J Rare Dis. 2017 Dec 7;12(1):177. doi: 10.1186/s13023-017-0730-1. PMID 29212508
- [Background] Bogart KR, Dermody SS. Relationship of rare disorder latent clusters to anxiety and depression symptoms. Health Psychol. 2020 Apr;39(4):307-315. doi: 10.1037/hea0000840. Epub 2019 Dec 19. PMID 31855040
- [Background] Rothrock NE, Amtmann D, Cook KF. Development and validation of an interpretive guide for PROMIS scores. J Patient Rep Outcomes. 2020 Feb 28;4(1):16. doi: 10.1186/s41687-020-0181-7. PMID 32112189
- [Background] Uhlenbusch N, Lowe B, Harter M, Schramm C, Weiler-Normann C, Depping MK. Depression and anxiety in patients with different rare chronic diseases: A cross-sectional study. PLoS One. 2019 Feb 20;14(2):e0211343. doi: 10.1371/journal.pone.0211343. eCollection 2019. PMID 30785907
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Saunders R, Moinian D, Stott J, Delamain H, Naqvi SA, Singh S, Wheatley J, Pilling S, Buckman JEJ. Measurement invariance of the PHQ-9 and GAD-7 across males and females seeking treatment for common mental health disorders. BMC Psychiatry. 2023 Apr 28;23(1):298. doi: 10.1186/s12888-023-04804-x. PMID 37118684
- [Background] Lai X, Jiang Y, Sun Y, Zhang Z, Wang S. Prevalence of depression and anxiety, and their relationship to social support among patients and family caregivers of rare bone diseases. Orphanet J Rare Dis. 2023 Jan 26;18(1):18. doi: 10.1186/s13023-022-02611-3. PMID 36703212
- [Background] Xiao SY. et al. The theoretical basis and applications of Social Support Rating Scale (SSRS). Journal of Clinical Psychiatry. 1994;4:98-100.
- [Background] Kenny T, et al. The importance of psychological support for parents and caregivers of children with a rare disease diagnosis. Rare Disease and Orphan Drugs Journal. 2022;1(2):7.
- [Background] Anderson M, Elliott EJ, Zurynski YA. Australian families living with rare disease: experiences of diagnosis, health services use and needs for psychosocial support. Orphanet J Rare Dis. 2013 Feb 11;8:22. doi: 10.1186/1750-1172-8-22. PMID 23398775
- [Background] Scharping M, Brennenstuhl H, Garbade SF, Wild B, Posset R, Zielonka M, Kolker S, Haun MW, Opladen T. Unmet Needs of Parents of Children with Urea Cycle Disorders. Children (Basel). 2022 May 12;9(5):712. doi: 10.3390/children9050712. PMID 35626889
- [Background] Lyon ME, Fraser JL, Thompkins JD, Clark H, Brodie N, Detwiler K, Torres C, Guerrera MF, Younge T, Aoun S, Trujillo Rivera EA. Advance Care Planning for Children With Rare Diseases: A Pilot RCT. Pediatrics. 2024 Jun 1;153(6):e2023064557. doi: 10.1542/peds.2023-064557. PMID 38699801
- [Background] Peterman AH, Fitchett G, Brady MJ, Hernandez L, Cella D. Measuring spiritual well-being in people with cancer: the functional assessment of chronic illness therapy--Spiritual Well-being Scale (FACIT-Sp). Ann Behav Med. 2002 Winter;24(1):49-58. doi: 10.1207/S15324796ABM2401_06. PMID 12008794
- [Background] Cooper B, Kinsella GJ, Picton C. Development and initial validation of a family appraisal of caregiving questionnaire for palliative care. Psychooncology. 2006 Jul;15(7):613-22. doi: 10.1002/pon.1001. PMID 16287207
- [Background] Toledano-Toledano F, Moral de la Rubia J, Dominguez-Guedea MT, Nabors LA, Barcelata-Eguiarte BE, Rocha-Perez E, Luna D, Leyva-Lopez A, Rivera-Rivera L. Validity and Reliability of the Beck Anxiety Inventory (BAI) for Family Caregivers of Children with Cancer. Int J Environ Res Public Health. 2020 Oct 23;17(21):7765. doi: 10.3390/ijerph17217765. PMID 33114144
- [Background] Alimujiang A, Wiensch A, Boss J, Fleischer NL, Mondul AM, McLean K, Mukherjee B, Pearce CL. Association Between Life Purpose and Mortality Among US Adults Older Than 50 Years. JAMA Netw Open. 2019 May 3;2(5):e194270. doi: 10.1001/jamanetworkopen.2019.4270. PMID 31125099
- [Background] Hill PL, Turiano NA. Purpose in life as a predictor of mortality across adulthood. Psychol Sci. 2014 Jul;25(7):1482-6. doi: 10.1177/0956797614531799. Epub 2014 May 8. PMID 24815612
- [Background] Boettcher J, Filter B, Denecke J, Hot A, Daubmann A, Zapf A, Wegscheider K, Zeidler J, von der Schulenburg JG, Bullinger M, Rassenhofer M, Schulte-Markwort M, Wiegand-Grefe S. Evaluation of two family-based intervention programs for children affected by rare disease and their families - research network (CARE-FAM-NET): study protocol for a rater-blinded, randomized, controlled, multicenter trial in a 2x2 factorial design. BMC Fam Pract. 2020 Nov 20;21(1):239. doi: 10.1186/s12875-020-01312-9. PMID 33218310
- [Background] First Michael B, et al. Structured Clinical Interview for DSM-IV-TR Axis I Disorders, Clinical Trials Version (SCID-CT). New York: Biometrics Research, New York State Psychiatric institute, 2007.
- [Background] Witt S, Schuett K, Wiegand-Grefe S, Boettcher J, Quitmann J. Living with a rare disease - experiences and needs in pediatric patients and their parents. Orphanet J Rare Dis. 2023 Aug 11;18(1):242. doi: 10.1186/s13023-023-02837-9. PMID 37568186
- [Background] Delisle VC, Gumuchian ST, Rice DB, Levis AW, Kloda LA, Korner A, Thombs BD. Perceived Benefits and Factors that Influence the Ability to Establish and Maintain Patient Support Groups in Rare Diseases: A Scoping Review. Patient. 2017 Jun;10(3):283-293. doi: 10.1007/s40271-016-0213-9. PMID 28004275
- [Background] Ashtari S, Taylor A. Patients With Rare Diseases and the Power of Online Support Groups: Implications for the Medical Community. JMIR Form Res. 2023 Sep 14;7:e41610. doi: 10.2196/41610. PMID 37707878
- [Background] Titgemeyer SC, Schaaf CP. Facebook Support Groups for Rare Pediatric Diseases: Quantitative Analysis. JMIR Pediatr Parent. 2020 Nov 19;3(2):e21694. doi: 10.2196/21694. PMID 33211019
- [Background] McCarthy SR, Golembiewski EH, Gravholt DL, Clark JE, Clark J, Fischer C, Mulholland H, Babcock K, Montori VM, Jones A. Documentation of Psychosocial Distress and Its Antecedents in Children with Rare or Life-Limiting Chronic Conditions. Children (Basel). 2022 May 5;9(5):664. doi: 10.3390/children9050664. PMID 35626841
- [Background] World Health Organization Group Problem Management Plus (Group PM+): group psychological help for adults impaired by distress in communities exposed to adversity. Generic field-trial version 1.0. 30 August 2020. https://www.who.int/publications/i/item/9789240008106
- [Background] Jordans MJD, Kohrt BA, Sangraula M, Turner EL, Wang X, Shrestha P, Ghimire R, Van't Hof E, Bryant RA, Dawson KS, Marahatta K, Luitel NP, van Ommeren M. Effectiveness of Group Problem Management Plus, a brief psychological intervention for adults affected by humanitarian disasters in Nepal: A cluster randomized controlled trial. PLoS Med. 2021 Jun 17;18(6):e1003621. doi: 10.1371/journal.pmed.1003621. eCollection 2021 Jun. PMID 34138875
- [Background] de Graaff AM, Cuijpers P, Twisk JWR, Kieft B, Hunaidy S, Elsawy M, Gorgis N, Bouman TK, Lommen MJJ, Acarturk C, Bryant R, Burchert S, Dawson KS, Fuhr DC, Hansen P, Jordans M, Knaevelsrud C, McDaid D, Morina N, Moergeli H, Park AL, Roberts B, Ventevogel P, Wiedemann N, Woodward A, Sijbrandij M; STRENGTHS Consortium; STRENGTHS consortium. Peer-provided psychological intervention for Syrian refugees: results of a randomised controlled trial on the effectiveness of Problem Management Plus. BMJ Ment Health. 2023 Feb;26(1):e300637. doi: 10.1136/bmjment-2022-300637. Epub 2023 Feb 8. PMID 36789918
- [Background] Weathers et al., The PTSD Checklist for DSM-5 (PCL-5) - Standard [Measurement instrument]. https://www.ptsd.va.gov
- [Background] Czachowski S, Seed P, Schofield P, Ashworth M. Measuring psychological change during cognitive behaviour therapy in primary care: a Polish study using 'PSYCHLOPS' (Psychological Outcome Profiles). PLoS One. 2011;6(12):e27378. doi: 10.1371/journal.pone.0027378. Epub 2011 Dec 15. PMID 22194783
- [Background] Ustun, et al. and World Health Organization. Measuring health and disability: manual for WHO Disability Assessment Schedule (WHODAS 2.0). World Health Organization 2010. Manual 16, June 2016.
- [Result] Ali AM, Schwalk DE, Lyon ME. Adapting and Beta Testing Rare Group Problem Management Plus for Family Caregivers of Children with Rare Diseases. (April 30, 2025). Poster. 2025 Awardee Medical Student Research Day, Abdulla Ali, in the category of Clinical and Translational Research. George Washington University School of Medicine and Health Sciences, Washington DC.